CLINICAL TRIAL: NCT05145010
Title: Phase 2, Open-Label, Long-Term, Extension (OLE) Study of Infigratinib, an FGFR 1-3-Selective Tyrosine Kinase Inhibitor, in Children With Achondroplasia: PROPEL OLE
Brief Title: Extension Study of Infigratinib in Children With Achondroplasia (ACH)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QBGJ398-203
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Achondroplasia
Keywords: Skeletal dysplasia; Endochondral ossification; Achondroplasia (ACH); Quality of life in achondroplasia; Fibroblast growth factor receptor 3; FGFR3; Endochondral bone formation; Short-limb disproportionate stature; Bone disease; Functionality in achondroplasia; Musculoskeletal diseases; Osteochondrodysplasia; Genetic diseases; Long - term treatment; Growth; Annualized height velocity; Treatment option; Tyrosine kinase inhibitor
MeSH Terms: conditions — Achondroplasia; Mucopolysaccharidosis IV; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Rollover subjects (Experimental): Children who have completed QED-sponsored interventional study with infigratinib (Phase 2 or Phase 3)
  Interventions: Drug: Infigratinib
- Arm 2: Treatment naïve subjects (Experimental): Children naïve to infigratinib
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Infigratinib minitablets or sprinkle capsules to be administered by mouth. In subjects that completed a prior study with infigratinib, the starting dose will be the same as the last dose received in the prior interventional study with infigratinib. Infigratinib dose may be adjusted to 0.25 mg/kg/day (the dose selected to be explored further in the dose escalation portion of Phase 2 study QBGJ398-201 (PROPEL 2)).
  Arms: Arm 1: Rollover subjects
Drug: Infigratinib — Infigratinib sprinkle capsules to be administered by mouth. Starting dose for the subjects naïve to Infigratinib will be 0.25 mg/kg/day (the dose selected to be explored further in the dose escalation portion of Phase 2 study QBGJ398-201 (PROPEL 2)).
  Arms: Arm 2: Treatment naïve subjects

SUMMARY:
This is a Phase 2, multicenter, open-label, extension (OLE) study to evaluate the long-term safety, tolerability, and efficacy of infigratinib, an FGFR 1-3-selective tyrosine kinase inhibitor, in subjects with ACH who previously completed a QED-sponsored interventional study, and potentially in additional subjects who are naïve to infigratinib treatment. Quality of Life assessments for this subject population will also be evaluated. Treatment-naïve subjects must have at least a 6-month period of growth assessment in study QBGJ398-001 (PROPEL) and will be enrolled in this OLE study only after a dose to be explored further is identified in Phase 2 Study QBGJ398-201 and subjects are not otherwise eligible to enroll in another QED-sponsored Phase 2 or Phase 3 ACH study.

ELIGIBILITY:
Key Rollover Subjects Inclusion Criteria:

1. Pediatric subjects with ACH who have completed a previous QED-sponsored interventional study with infigratinib.
2. Subjects and parent(s), legal guardian(s), or caregiver(s) are willing and able to comply with study visits and study procedures.
3. Subjects are able to swallow oral medication.
4. Negative pregnancy test in girls ≥10 years of age or girls of any age who have experienced menarche.
5. If sexually active, subject must be willing to use a highly effective method of contraception while taking study drug and for 1 month after the last dose of study drug.
6. The PI, or a person designated by the PI, will obtain written informed consent from each subject's parent(s), legal guardian(s), or caregiver(s) and the subject's assent, when applicable, before any study-specific activity is performed.

Key Rollover Subjects Exclusion Criteria:

1. Subject has concurrent circumstance, disease, or condition that, in the view of the PI and/or sponsor, would interfere with study participation or safety evaluations.
2. Subjects who developed a medical condition that will require the initiation of treatment with a prohibited medication.
3. Subjects prematurely discontinued a prior QED-sponsored interventional study with infigratinib
4. Current participation in an ongoing clinical study with a sponsor other than QED
5. Subjects that have reached final height or near final height.

Key Inclusion Criteria for Treatment Naïve Subjects

1. Subject must be 3 to <18 years of age at screening and have growth potential.
2. Subjects and parent(s), legal guardian(s), or caregiver(s) are willing and able to comply with study visits and study procedures.
3. Subjects are able to swallow oral medication.
4. Subjects who have a diagnosis of ACH, documented clinically and confirmed by genetic testing.
5. Subjects have at least a 6-month period of growth assessment in the PROPEL study (Protocol QBGJ398 001) before study entry.
6. Negative pregnancy test in girls ≥10 years of age or girls of any age who have experienced menarche.
7. If sexually active, subject must be willing to use a highly effective method of contraception while taking study drug and for 1 month after the last dose of study drug.
8. The PI, or a person designated by the PI, will obtain written informed consent from each subject's parent(s), legal guardian(s), or caregiver(s) and the subject's assent, when applicable, before any study-specific activity is performed.

Key Exclusion Criteria for Treatment Naïve Subjects

1. Subjects who have hypochondroplasia or short stature condition other than ACH (e.g., trisomy 21, pseudoachondroplasia, psychosocial short stature).
2. Subjects who have significant concurrent disease or condition that, in the view of the PI and/or sponsor, would represent an increased risk to the subject or would interfere with study participation or safety evaluations.
3. Subjects who have a history of malignancy.
4. Subjects who are currently receiving treatment with agents that are known strong inducers or inhibitors of cytochrome P450 (CYP) 3A4.
5. Subjects who discontinued treatment with prohibited medications for at least 5 half-lives before screening are eligible.
6. Subjects who have received treatment with growth hormone, insulin-like growth factor 1 (IGF 1), anabolic steroids or any investigational or approved drug for the treatment of ACH in the previous 6 months.
7. Subjects who have significant abnormality in screening laboratory results.
8. Subjects who have had a fracture within 12 months of screening.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2031-12-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAE) and serious TEAE | 10 years
Changes over time in height Z-score in relation to ACH and non-ACH growth charts | 10 years

SECONDARY OUTCOMES:
Changes over time in absolute height velocity, expressed as height velocity Z-score in relation to ACH and non ACH growth charts | 10 years
Changes over time in body proportions | 10 years
Changes over time in weight z-score | 10 years
Changes overtime in BMI | 10 years
Age of puberty onset and time to Tanner stage ≥4 | 10 years
Changes over time in number of episodes of otitis media per year | 10 years
Changes over time in number of episodes and/or severity of sleep apnea | 10 years
Changes over time in range of motion (elbow) | 10 years
Changes over time in skeletal abnormalities of the lower extremities and spine | 10 years
Changes in health-related Quality of life [HRQoL] as assessed by Pediatric Quality of Life Inventory (PedsQL) | 10 years
Changes in health-related Quality of life [HRQoL] as assessed by Quality of Life in Short Stature Youth questionnaire (QoLISSY) | 10 years
Overall pain as assessed by Numeric Rating Scale for pain (Pain-NRS) | 10 years
Changes in functional abilities as evaluated by Functional Independence Measure for Children (WeeFIM) | 10 years
Severity of the physical functioning challenges as assessed by Patient/Parent Global Impression of Severity (PGI-S) | 10 years
Severity of the physical functioning challenges as assessed by Patient/Parent Global Impression of Change (PGI-C) | 10 years
Subject and caregiver evaluation of treatment benefit as assessed by a qualitative interview | 10 years
Changes in cognitive functions assessed by age-appropriate computerized tests | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: QED Therapeutics SVP, Clinical Development, Study Director — QED Therapeutics
Locations (31):
- United States (8):
  - USCF Benioff Children's Hospital, Oakland, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins University, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Hospital de Pediatría SAMIC Prof. Dr. Juan P. Garrahan, Ciudad Autonoma Buenos Aires, Buenos Aires, Argentina
- Murdoch Children's Hospital, Parkville, Victoria, Australia
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (3):
  - Hopital Femme Mere Enfant, Lyon
  - Hopital Necker-Enfants Malades, Paris
  - Hopital des Enfants, Toulouse
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Policlinico A. Gemelli IRCCS, Roma
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- KK Women's and Children's Hosptial, Singapore, Singapore
- Spain (3):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Vithas San José, Vitoria-Gasteiz, Álava
- United Kingdom (6):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - St. Thomas' Hospital, London
  - Manchester University Children's Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No